CLINICAL TRIAL: NCT07224555
Title: Pilot Study to Evaluate the Efficacy and Safety of Xtressé™ Gummy-Based Nutraceutical Supplement in Women With Self-Perceived Thinning Hair
Brief Title: Study Evaluating Xtressé Gummy Supplement in Women With Self-Perceived Thinning Hair
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Restore Biologics Holdings, Inc. dba Xtressé (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XTS-2025-001
Record Dates: First submitted 2025-10-29; First posted 2025-11-04 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Hair Thinning
Keywords: hair loss; thin hair; thinning hair; Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Intervention Model Description: Open label study evaluating safety and efficacy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Xtressé Nutraceutical Supplement Active (Experimental): Other: Xtressé Nutraceutical Supplement Participants will receive a 30 day supply of gummy supplement 4 times during the study. Participants will take supplement daily and notate usage in log.
  Interventions: Other: Xtressé Hair Growth Gummies

INTERVENTIONS:
Other: Xtressé Hair Growth Gummies — The nutraceutical supplement is powered by proprietary X-3 BioActive Blend and contains plant based extracts and regenerative compounds not commonly found in existing hair supplements.

SUMMARY:
The goal of this study is to determine how safe and effective it is to improve hair growth using an active gummy treatment in women with self-perceived thinning hair.

The main aims of this trial are:

1. To confirm using photographic analysis, changes in the quality, volume, and thickness of hair.
2. To gauge patient satisfaction with hair changes and application process.
3. Monitor and report any adverse events associated with the daily intake of Xtressé

Participants who qualify will complete 5 visits after voluntary consent has been given. Participants will be given a 30-day supply of the gummies at each visit over a 4-month period. Photographs and scalp analysis will be performed at each visit to measure changes in hair volume, thickness, and growth.

DETAILED DESCRIPTION:
In the study, participants will be asked to complete the following:

* Provide basic personal information (including date of birth, gender, race and ethnicity)
* Provide their medical/ surgical history and perform a medical exam (including but not limited to symptom-directed physical exam, skin type, vital signs, height, weight, and pregnancy test)
* Follow study rules such as avoiding certain medications and treatments
* Provide information on any medications, treatments or reactions that started after the study began
* Take gummy treatment daily and complete a treatment diary
* Allow clinical assessments and documentation of the treatment, such as photography, hair density measurements, any reactions or side effects

To qualify for this trial, participants must:

* Be a female adult between 28 to 65 years of age
* Have consistent self-perceived thinning hair.
* Give voluntary written consent
* Be willing to follow study instructions and complete study requirements, including maintaining current diet and hair care routine, not using non-approved lotions and creams on the treatments areas
* Allow photographs of the front and top area of the scalp
* Not be pregnant or breast feeding before and during the study and agree to use acceptable forms of birth control
* Confirm they are not sensitive to any of the study treatment ingredients

All photographs of the treatment area collected during the study will be used as study data.

All participants have the right to refuse further participation in the study at any time.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-65 years with self-perceived thinning hair (confirmed by an investigator).
* Fitzpatrick skin types I to VI.
* Ability and willingness to comply with the study protocol.
* Commitment to using effective contraception throughout the study if of childbearing potential.

Exclusion Criteria:

* Pregnancy, nursing, or recent initiation of hormone therapy.
* Change in other hair treatments within 3 months prior to the study.
* Known uncontrolled health conditions (e.g., poorly controlled diabetes, hypertension).
* History of hair or scalp disorders that could interfere with study results.
* History of metabolic syndrome.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female sex at birth
Enrollment: 60 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Hair Density Changes measured by SOCAi | From enrollment to the end of the study at 4 months
  Images will be captured using the the SOCAi system at baseline and Days 30, 60, 90, and 120, to evaluate hair density changes.
Within-subject increase in hair density assessed via Canfield HairMetrix® Phototrichogram Analysis | From enrollment to the end of treatment at 4 months
  Quantitative hair measurements calculated by analyzing the participants digital images from baseline to 4 months after taking Xtressé™ Supplements. Measurements of density as measured hair per cm².
Within-subject increase in hair thickness assessed via Canfield HairMetrix® Phototrichogram Analysis | From enrollment to the end of treatment at 4 months
  Quantitative hair measurements calculated by analyzing the participants digital images from baseline to 4 months after taking Xtressé™ Supplements. Measurements of follicular unit vellus/terminal ratio.

SECONDARY OUTCOMES:
Incidence of Adverse Events associated with Treatment | From first treatment until the end of treatment at 4 months
  Collect and quantify the incidence of treatment-related adverse events and treatment-related serious adverse events associated with the daily intake of supplement

OTHER OUTCOMES:
Participant self-assessment of hair improvements collected via questionnaire | From enrollment to the end of study at 4 months
  Observations and changes noted in hair loss graded on scale of 0 to 4 with 0 as no change and 4 as a very severe outcome.
  Observations and changes noted in quality of life based on hair loss, with outcomes graded between extremely effected to not at all.
  Observations are based on self-assessments completed at baseline and Day 120.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Y Rayner, MS, Study Director — Restore Biologics Holdings, Inc. dba Xtressé
Locations (4):
- United States (4):
  - Advanced Dermatology & Cosmetic Surgery, Maitland, Florida
  - Hair Medicine Institute, Alpharetta, Georgia
  - Kindred Hair and Skin, Marriottsville, Maryland
  - Root Hair Institute, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No